CLINICAL TRIAL: NCT01601704
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Assessing the Occurrence of Major Adverse Cardiovascular Events (MACE) in Overweight and Obese Subjects With Cardiovascular Risk Factors Receiving Naltrexone SR/Bupropion SR
Brief Title: Cardiovascular Outcomes Study of Naltrexone SR/Bupropion SR in Overweight and Obese Subjects With Cardiovascular Risk Factors (The Light Study)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NB-CVOT; The Light Study (Other: Takeda); U1111-1162-4981 (Registry Identifier: WHO)
Record Dates: First submitted 2012-05-14; First posted 2012-05-18 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2016-04

CONDITIONS: Obesity; Overweight
Keywords: Body Weight; Bupropion; Cardiovascular Diseases; Diabetes Mellitus; Diabetes Mellitus, Type 2; Endocrine System Diseases; Glucose Metabolism Disorders; Heart Diseases; Metabolic Diseases; Narcotic Antagonists; Naltrexone; Nutrition Disorders; Obesity; Overnutrition; Overweight
MeSH Terms: conditions — Obesity; Overweight; Body Weight; Cardiovascular Diseases; Diabetes Mellitus; Diabetes Mellitus, Type 2; Endocrine System Diseases; Glucose Metabolism Disorders; Heart Diseases; Metabolic Diseases; Nutrition Disorders; Overnutrition | interventions — bupropion hydrochloride, naltrexone hydrochoride drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NB32 (Experimental)
  Interventions: Drug: NB32; Behavioral: Weight Management Program
- PBO (Placebo Comparator)
  Interventions: Drug: PBO; Behavioral: Weight Management Program

INTERVENTIONS:
Drug: NB32 — Naltrexone SR 32 mg/Bupropion SR 360 mg/day. Administered in addition to the weight management program.
  Other Names: CONTRAVE
  Arms: NB32
Drug: PBO — Placebo. Administered in addition to the weight management program.
  Arms: PBO
Behavioral: Weight Management Program — A comprehensive weight management program will be administered in addition to the subject's study medication assignment. The program includes internet counseling by an accredited health and fitness professional and a nutrition and exercise program with goal setting and educational and tracking tools.
  Other Names: WeightMate (Tm)

SUMMARY:
The purpose of this study is to determine the effects of NB relative to placebo on major adverse cardiovascular events (MACE) such as cardiovascular death, non-fatal myocardial infarction, and non-fatal stroke in overweight and obese subjects who are at a higher risk of having these events because they have diabetes and/or other cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. ≥50 years of age (women) or ≥45 years of age (men)
2. Body mass index (BMI) ≥27 kg/m2 and ≤50 kg/m2
3. Waist circumference ≥88 cm (women) or ≥102 cm (men)
4. At increased risk of adverse cardiovascular outcomes:

   * Cardiovascular disease (confirmed diagnosis or at high likelihood of cardiovascular disease) with at least one of the following:

     * History of documented myocardial infarction >3 months prior to screening
     * History of coronary revascularization
     * History of carotid or peripheral revascularization
     * Angina with ischemic changes (resting ECG), ECG changes on a graded exercise test (GXT), or positive cardiac imaging study
     * Ankle brachial index <0.9 (by simple palpation) within prior 2 years
     * ≥50% stenosis of a coronary, carotid, or lower extremity artery within prior 2 years

AND/OR

* Type 2 diabetes mellitus with at least 2 of the following:

  * Hypertension (controlled with or without pharmacotherapy at <145/95 mm Hg)
  * Dyslipidemia requiring pharmacotherapy
  * Documented low HDL cholesterol (<50 mg/dL in women or <40 mg/dL in men) within prior 12 months
  * Current tobacco smoker

Exclusion Criteria:

1. Myocardial infarction within 3 months prior to screening
2. Angina pectoris Grade III or IV as per the Canadian Cardiovascular Society grading scheme
3. Clinical history of cerebrovascular disease (stroke)
4. History of tachyarrhythmia other than sinus tachycardia
5. Planned bariatric surgery, cardiac surgery, or coronary angioplasty
6. History of seizures (including febrile seizures), cranial trauma, or other conditions that predispose the subject to seizures
7. History of mania or current diagnosis of active psychosis, active bulimia or anorexia nervosa (binge eating disorder is not exclusionary)
8. Any condition with life expectancy anticipated to be less than 4 years (e.g., congestive heart failure NYHA Class 3 or 4)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8910 (Actual)
Dates: Start 2012-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (224):
- United States (224):
  - Birmingham, Alabama
  - Dothan, Alabama
  - Mobile, Alabama
  - Scottsboro, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Peoria, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Tuscson, Arizona
  - Little Rock, Arkansas
  - Anaheim, California
  - Carmichael, California
  - Escondido, California
  - Fresno, California
  - Harbor City, California
  - Huntington Beach, California
  - La Jolla, California
  - Lomita, California
  - Los Angeles, California
  - Paramount, California
  - Pasadena, California
  - Riverside, California
  - Sacramento, California
  - Santa Rosa, California
  - Spring Valley, California
  - Thousand Oaks, California
  - Torrance, California
  - West Hills, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Golden, Colorado
  - Wheat Ridge, Colorado
  - Norwalk, Connecticut
  - Stamford, Connecticut
  - Wilmington, Delaware
  - Washington D.C., District of Columbia
  - Boynton Beach, Florida
  - Brooksville, Florida
  - Clearwater, Florida
  - DeLand, Florida
  - Delray Beach, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Jacksonville Beach, Florida
  - Melbourne, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - New Smyrna Beach, Florida
  - Oakland Park, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Pembroke Pines, Florida
  - Pensacola, Florida
  - Pinellas Park, Florida
  - St. Petersburg, Florida
  - Vero Beach, Florida
  - Wellington, Florida
  - Winter Haven, Florida
  - Atlanta, Georgia
  - Austell, Georgia
  - Columbus, Georgia
  - Lawrenceville, Georgia
  - Riverdale, Georgia
  - Savannah, Georgia
  - Stockbridge, Georgia
  - Honolulu, Hawaii
  - Meridian, Idaho
  - Chicago, Illinois
  - Gurnee, Illinois
  - Melrose Park, Illinois
  - Bloomington, Indiana
  - Brownsburg, Indiana
  - Elwood, Indiana
  - Evansville, Indiana
  - Hammond, Indiana
  - South Bend, Indiana
  - Valparaiso, Indiana
  - Ames, Iowa
  - Council Bluffs, Iowa
  - Des Moines, Iowa
  - West Des Moines, Iowa
  - Overland Park, Kansas
  - Wichita, Kansas
  - Crestview Hills, Kentucky
  - Louisville, Kentucky
  - Mount Sterling, Kentucky
  - Alexandria, Louisiana
  - Baton Rouge, Louisiana
  - Monroe, Louisiana
  - Natchitoches, Louisiana
  - Auburn, Maine
  - Bangor, Maine
  - Baltimore, Maryland
  - Columbia, Maryland
  - Elkridge, Maryland
  - Lutherville, Maryland
  - Salisbury, Maryland
  - Boston, Massachusetts
  - Brockton, Massachusetts
  - Fall River, Massachusetts
  - Haverhill, Massachusetts
  - Methuen, Massachusetts
  - Bingham Farms, Michigan
  - Dearbon, Michigan
  - Kalamazoo, Michigan
  - Midland, Michigan
  - Saginaw, Michigan
  - Southfield, Michigan
  - Stevensville, Michigan
  - Edina, Minnesota
  - Rochester, Minnesota
  - Jackson, Mississippi
  - Olive Branch, Mississippi
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Butte, Montana
  - Missoula, Montana
  - Fremont, Nebraska
  - Grand Island, Nebraska
  - Omaha, Nebraska
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Reno, Nevada
  - Sparks, Nevada
  - Belvidere, New Jersey
  - Edison, New Jersey
  - Elizabeth, New Jersey
  - Elmer, New Jersey
  - Linden, New Jersey
  - Ridgewood, New Jersey
  - Albuquerque, New Mexico
  - Endwell, New York
  - New Hyde Park, New York
  - New York, New York
  - Staten Island, New York
  - Syracuse, New York
  - The Bronx, New York
  - Williamsville, New York
  - Cary, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Elizabeth City, North Carolina
  - Greensboro, North Carolina
  - Greenville, North Carolina
  - Hickory, North Carolina
  - Morganton, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Beachwood, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Delaware, Ohio
  - Kettering, Ohio
  - Marion, Ohio
  - Mentor, Ohio
  - Willoughby Hills, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Altoona, Pennsylvania
  - Bensalem, Pennsylvania
  - Danville, Pennsylvania
  - Duncansville, Pennsylvania
  - Ephrata, Pennsylvania
  - Jersey Shore, Pennsylvania
  - Lancaster, Pennsylvania
  - Lansdale, Pennsylvania
  - Norristown, Pennsylvania
  - Scottdale, Pennsylvania
  - Sellersville, Pennsylvania
  - State College, Pennsylvania
  - West Reading, Pennsylvania
  - Wilkes-Barre, Pennsylvania
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Greer, South Carolina
  - Hodges, South Carolina
  - Laurens, South Carolina
  - Mt. Pleasant, South Carolina
  - Rapid City, South Dakota
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Jackson, Tennessee
  - Kingsport, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Beaumont, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - Hurst, Texas
  - Lake Jackson, Texas
  - McKinney, Texas
  - San Antonio, Texas
  - Schertz, Texas
  - Tomball, Texas
  - Waco, Texas
  - Bountiful, Utah
  - Draper, Utah
  - Murray, Utah
  - Ogden, Utah
  - Orem, Utah
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Alexandria, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Winchester, Virginia
  - Seattle, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Walla Walla, Washington
  - Green Bay, Wisconsin
  - Kenosha, Wisconsin
  - Madison, Wisconsin

REFERENCES:
- [Derived] Nissen SE, Wolski KE, Prcela L, Wadden T, Buse JB, Bakris G, Perez A, Smith SR. Effect of Naltrexone-Bupropion on Major Adverse Cardiovascular Events in Overweight and Obese Patients With Cardiovascular Risk Factors: A Randomized Clinical Trial. JAMA. 2016 Mar 8;315(10):990-1004. doi: 10.1001/jama.2016.1558. PMID 26954408

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Administered in addition to the weight management program.
  Weight Management Program: A comprehensive weight management program will be administered in addition to the subject's study medication assignment. The program includes internet counseling by an accredited health and fitness professional and a nutrition and exercise program with goal setting and educational and tracking tools.
Period: Overall Study
Arm/Group | NB32 | Placebo
Started (Represents number of participants randomized) | 4456 | 4454
Treated (Represents number of participants included in the ITT analysis) | 4455 | 4450
Completed (Completed indicates treated participants. Represents number of participants in the ITT analysis.) | 4455 | 4450
Not Completed | 1 | 4
Not completed — Randomized but not dispensed study med | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NB32 | Placebo | Total
Number analyzed (Participants) | 4455 | 4450 | 8905
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2973 | 3053 | 6026
  >=65 years | 1482 | 1397 | 2879
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (7.27) | 60.9 (7.38) | 61.0 (7.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2437 | 2419 | 4856
  Male | 2018 | 2031 | 4049
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 279 | 291 | 570
  Not Hispanic or Latino | 4174 | 4156 | 8330
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 20 | 31
  Asian | 19 | 27 | 46
  Native Hawaiian or Other Pacific Islander | 6 | 6 | 12
  Black or African American | 656 | 648 | 1304
  White | 3738 | 3698 | 7436
  More than one race | NA — Selection of multiple race categories was not permissible by the participants. Participants advised to select the most appropriate category. | NA — Selection of multiple race categories was not permissible by the participants. Participants advised to select the most appropriate category. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 25 | 51 | 76
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4455 | 4450 | 8905
Weight [Mean (Standard Deviation); unit: kilogram] | 105.6 (19.09) | 106.3 (19.18) | 106.0 (19.14)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI was calculated at the site. Data are missing for 3 participants for whom the site did not calculate BMI, although weight and height were measured.
  kg/m^2
    number analyzed (Participants) | 4452 | 4450 | 8902
    (all) | 37.2 (5.26) | 37.4 (5.44) | 37.3 (5.35)
Cardiovascular (CV) risk group [Count of Participants; unit: Participants]
  CV disease without T2DM (type 2 diabetes mellitus) | 670 | 646 | 1316
  CV disease with T2DM | 745 | 801 | 1546
  T2DM without CV disease | 3039 | 3002 | 6041
Hypertension [Count of Participants; unit: Participants]
  Yes | 4162 | 4117 | 8279
  No | 293 | 333 | 626
Dyslipidemia [Count of Participants; unit: Participants]
  Yes | 4100 | 4070 | 8170
  No | 355 | 380 | 735
History of Depression [Count of Participants; unit: Participants]
  Yes | 1031 | 995 | 2026
  No | 3424 | 3455 | 6879
Baseline Antidepressant Medication Use [Count of Participants; unit: Participants] | 1042 | 1015 | 2057

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Confirmed Occurrence of Major Adverse Cardiovascular Event (MACE)
Description: The primary endpoint is the time from randomization to the first confirmed occurrence of any event within the primary MACE composite (defined as cardiovascular death, nonfatal myocardial infarction, or nonfatal stroke). Due to early termination of the study, pre-planned 50% interim analysis is considered the primary analysis for outcome measures. The pre-planned 50% interim analysis was conducted when 50% of the total planned MACE were observed.
Time Frame: Confirmed occurrence of event between Day 1 (randomization) and up to a maximum of 4 years of follow-up
Population: Intent-to-treat (ITT) population is defined as subjects who undergo randomization into the Treatment Period (TP) and are dispensed study medication. Treatment refers to the treatment assigned during TP randomization rather than the actual treatment received. ITT population is the primary analysis population for the primary and secondary endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 4455 | 4450
Participants | 90 | 102
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Non-Inferiority or Equivalence — At the pre-planned 50% interim analysis, a non-inferiority analysis was conducted based on the estimated hazard ratio (NB32/Placebo) for the time to the first confirmed occurrence of MACE. The upper-bound of the 99.7% confidence interval for the hazard ratio was compared to 1.4, the non-inferiority margin; Cox Proportional Hazard = 0.88, 99.7% CI 2-sided [0.57 to 1.34] — Hazard ratio is based on CPH model with treatment as a factor

2. Secondary Outcome: Percentage of Participants With a Confirmed Occurrence of Cardiovascular Death, Nonfatal Myocardial Infarction, Nonfatal Stroke, or Nonfatal Unstable Angina Requiring Hospitalization
Description: Due to early termination of the study, the pre-planned 50% interim analysis is considered the primary analysis for outcome measures.
Time Frame: Confirmed occurrence of event between Day 1 (randomization) and up to a maximum of 4 years of follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 4455 | 4450
Participants | 133 | 142
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; Cox Proportional Hazard = 0.93, 99.7% CI 2-sided [0.66 to 1.33] — Hazard ratio is based on CPH model with treatment as a factor

3. Secondary Outcome: Percentage of Participants With a Confirmed Occurrence of Cardiovascular Death (Including Fatal Myocardial Infarction, Fatal Stroke)
Description: as for outcome 2
Time Frame: Confirmed occurrence of event between Day 1 (randomization) and up to a maximum of 4 years of follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 4455 | 4450
Participants | 17 | 34
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; Cox Proportional Hazard = 0.50, 99.7% CI 2-sided [0.21 to 1.19] — Hazard ratio is based on CPH model with treatment as a factor

4. Secondary Outcome: Percentage of Participants With a Confirmed Occurrence of Myocardial Infarction (Nonfatal or Fatal)
Description: as for outcome 2
Time Frame: Confirmed occurrence of event between Day 1 (randomization) and up to a maximum of 4 years of follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 4455 | 4450
Participants | 55 | 57
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; Cox Proportional Hazard = 0.96, 99.7% CI 2-sided [0.55 to 1.67] — Hazard ratio is based on CPH model with treatment as a factor

5. Secondary Outcome: Percentage of Participants With a Confirmed Occurrence of Stroke (Nonfatal or Fatal)
Description: as for outcome 2
Time Frame: Confirmed occurrence of event between Day 1 (randomization) and up to a maximum of 4 years of follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 4455 | 4450
Participants | 22 | 21
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; Cox Proportional Hazard = 1.04, 99.7% CI 2-sided [0.43 to 2.55] — Hazard ratio is based on CPH model with treatment as a factor

ADVERSE EVENTS:
Time Frame: Treatment-emergent serious adverse events and treatment-emergent adverse events leading to study medication discontinuation are defined as those events with onset coincident with treatment period randomization starting at Visit 3 (Day 1) and through end of study or 30 days after discontinuation of study medication (whichever one is earlier).
Description: Safety data is based on all available data at the time of database lock, which occurred after the pre-planned 50% interim analysis.
Arm/Group | NB32 | Placebo
Serious Adverse Events (participants affected / at risk) | 463/4455 | 386/4450
Other Adverse Events (participants affected / at risk) | 1157/4455 | 282/4450
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NB32 (N=4455) | Placebo (N=4450)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Accelerated idioventricular rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 4 (6) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 11 (11) | 7 (7)
Angina pectoris (Cardiac disorders) | 17 (17) | 15 (15)
Angina unstable (Cardiac disorders) | 22 (25) | 15 (16)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 12 (12) | 15 (15)
Atrial flutter (Cardiac disorders) | 4 (5) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (3) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 13 (16) | 8 (11)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 2 (2)
Chronotropic incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 21 (22) | 21 (21)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 5 (5)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial infarction (Cardiac disorders) | 14 (14) | 13 (13)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 2 (2) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 3 (3) | 2 (2)
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Porphyria acute (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hiatus hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 4 (4)
Pancreatitis acute (Gastrointestinal disorders) | 3 (3) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 9 (10) | 3 (5)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 15 (15) | 9 (9)
Cyst (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 4 (4) | 2 (2)
Device dislocation (General disorders) | 1 (1) | 1 (1)
Device malfunction (General disorders) | 1 (1) | 0 (0)
Fat tissue increased (General disorders) | 0 (0) | 1 (1)
Ischaemic ulcer (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 22 (22) | 13 (13)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1)
Surgical failure (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 1 (1)
Unevaluable event (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 4 (4)
Cholecystitis acute (Hepatobiliary disorders) | 4 (4) | 5 (5)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 2 (2)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 2 (2)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 3 (3)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Bursitis infective staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 16 (17) | 8 (8)
Cellulitis of male external genital organ (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Colonic abscess (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 3 (3) | 6 (7)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (5) | 2 (2)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Human ehrlichiosis (Infections and infestations) | 1 (1) | 0 (0)
Infected bites (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 3 (3) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 12 (13) | 10 (10)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 5 (5)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Wound abscess (Infections and infestations) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal cord injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anticoagulation drug level below therapeutic (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 2 (2) | 0 (0)
Thyroid function test abnormal (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Alkalosis hypochloraemic (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 8 (9) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 40 (42) | 41 (44)
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Resorption bone increased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell unclassifiable lymphoma high grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 5 (5)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian granulosa cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (6)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem stroke (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery disease (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 2 (2) | 2 (2)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 7 (7) | 5 (5)
Complicated migraine (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Dementia with Lewy bodies (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic hyperosmolar coma (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Lacunar infarction (Nervous system disorders) | 2 (2) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Nerve root compression (Nervous system disorders) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Spondylitic myelopathy (Nervous system disorders) | 2 (2) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 7 (7) | 6 (6)
Transient ischaemic attack (Nervous system disorders) | 2 (3) | 4 (4)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 2 (2)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 3 (3) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 4 (4)
Nephrosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 8 (8) | 11 (11)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Endometrial hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Ovarian mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Gastrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 2 (2)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 1 (1)
Haematoma (Vascular disorders) | 2 (2) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 4 (4)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 3 (3) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NB32 (N=4455) | Placebo (N=4450)
Angina pectoris (Cardiac disorders) | 4 (4) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac discomfort (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac flutter (Cardiac disorders) | 2 (2) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 20 (20) | 5 (5)
Tachycardia (Cardiac disorders) | 3 (3) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 5 (5) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 11 (11) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 27 (27) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 18 (18) | 6 (6)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 18 (18) | 4 (4)
Bowel movement irregularity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 129 (129) | 15 (15)
Diarrhoea (Gastrointestinal disorders) | 35 (35) | 21 (21)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 21 (21) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 12 (12) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (3) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 3 (3)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 2 (2) | 2 (2)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 346 (346) | 21 (21)
Oesophageal rupture (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 3 (3) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 89 (89) | 1 (1)
Vomiting projectile (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 2 (2)
Chest discomfort (General disorders) | 2 (2) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Drug intolerance (General disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 13 (13) | 1 (1)
Feeling abnormal (General disorders) | 7 (7) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 0 (0)
Feeling jittery (General disorders) | 16 (16) | 1 (1)
Feeling of body temperature change (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 3 (3) | 0 (0)
Local swelling (General disorders) | 0 (0) | 1 (1)
Mucosal dryness (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 4 (4) | 1 (1)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 20 (20) | 14 (14)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0)
Grip strength decreased (Investigations) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 2 (2) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperphagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 11 (11)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 3 (3) | 4 (4)
Balance disorder (Nervous system disorders) | 2 (2) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 7 (7) | 2 (2)
Dizziness (Nervous system disorders) | 64 (67) | 8 (8)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 16 (16) | 0 (0)
Dysgraphia (Nervous system disorders) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0)
Essential tremor (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 51 (51) | 15 (15)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 4 (4) | 2 (2)
Memory impairment (Nervous system disorders) | 3 (3) | 4 (4)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 1 (1)
Muscle contractions involuntary (Nervous system disorders) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Neurodegenerative disorder (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 2 (2)
Spinal meningeal cyst (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 80 (81) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 5 (5) | 0 (0)
Affect lability (Psychiatric disorders) | 3 (3) | 3 (3)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1)
Anger (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 26 (26) | 8 (8)
Apathy (Psychiatric disorders) | 1 (1) | 0 (0)
Aversion (Psychiatric disorders) | 1 (1) | 0 (0)
Bruxism (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 5 (5) | 2 (2)
Depression (Psychiatric disorders) | 5 (5) | 10 (10)
Disorientation (Psychiatric disorders) | 4 (4) | 0 (0)
Fear (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 10 (10) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 2 (2) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 38 (38) | 16 (16)
Irritability (Psychiatric disorders) | 7 (7) | 2 (2)
Libido decreased (Psychiatric disorders) | 2 (2) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Middle insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Mood altered (Psychiatric disorders) | 2 (2) | 0 (0)
Mood swings (Psychiatric disorders) | 1 (1) | 1 (1)
Nervousness (Psychiatric disorders) | 8 (8) | 0 (0)
Nightmare (Psychiatric disorders) | 6 (6) | 2 (2)
Obsessive-compulsive disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 2 (2) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0)
Psychomotor retardation (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Sleep talking (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep terror (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ejaculation disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 3 (3)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 10 (10) | 3 (3)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
Cardioversion (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 3 (3) | 1 (1)
Hot flush (Vascular disorders) | 10 (10) | 2 (2)
Hypertension (Vascular disorders) | 25 (25) | 11 (11)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Labile blood pressure (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early. Outcome measures data is based on the 50% interim analysis, designated as the primary analysis. Safety data is based on all available data at the time of database lock, which occurred after the 50% interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If not already published by Sponsor as part of a multi-center publication, 24 months after conclusion, abandonment or termination of the study or notification that there will be no such multi-center publication, PI may publish the results for PI's study center individually. Prior to such publication, PI must provide Sponsor with at least 90 days to review and comment on the proposed publication. Sponsor may delay publication for up to an additional 6-month period to file for patent protection.